CLINICAL TRIAL: NCT04318795
Title: Minimally Invasive Spinal Decompression (MIS-D) Versus Minimally Invasive Spinal Decompression and Fusion (MIS-TLIF) for the Treatment of Lumbar Spinal Stenosis (LSS): A Prospective Randomized Controlled Trial
Brief Title: MIS-D Versus MIS-TLIF for the Treatment of Lumbar Spinal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Limin Rong, Prof., M.D., Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIS-D V.s. MIS-TLIF for LSS
Record Dates: First submitted 2020-03-16; First posted 2020-03-24 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Spinal Stenosis
Keywords: lumbar spinal stenosis; minimally invasive spine surgery; decompression; fusion; randomized controlled trial
MeSH Terms: conditions — Spinal Stenosis | interventions — Gene Fusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- minimally invasive spinal decompression (MIS-D) (Experimental): lumbar spinal decompression alone using minimally invasive approach, without any fusion or implantation
  Interventions: Procedure: minimally invasive spinal decompression (MIS-D)
- minimally invasive spinal decompression and fusion (MIS-TLIF) (Experimental): lumbar spinal decompression plus interbody fusion with implantation using minimally invasive approach
  Interventions: Procedure: minimally invasive spinal decompression and fusion (MIS-TLIF)

INTERVENTIONS:
Procedure: minimally invasive spinal decompression (MIS-D) — lumbar spinal decompression alone using minimally invasive approach, without any fusion or implantation
  Arms: minimally invasive spinal decompression (MIS-D)
Procedure: minimally invasive spinal decompression and fusion (MIS-TLIF) — lumbar spinal decompression plus interbody fusion with implantation using minimally invasive approach
  Arms: minimally invasive spinal decompression and fusion (MIS-TLIF)

SUMMARY:
The purpose of this study is to evaluate the effectiveness of two minimal invasive spine surgery, minimally invasive spinal decompression (MIS-D) and minimally invasive spinal decompression and fusion (MIS-TLIF), for patients diagnosed with lumbar spinal stenosis in terms of clinical outcomes, complications, reoperations, and other perioperative data.

DETAILED DESCRIPTION:
Lumbar spinal stenosis (LSS) is one of the most common degenerative spine diseases in older people and is associated with mechanical low back pain, radiculopathy and/or neurological claudication. The results of The Spine Patient Outcomes Research Trial (SPORT) reported that, surgical treatment in these patients led to significantly greater improvement in pain and function than nonsurgical treatment. Nowadays, decompression with instrumented or non-instrumented fusion is commonly practiced which is regarded as the "gold standard" surgery for LSS.

Over the last two decades, several retrospective studies comparing the surgical outcomes of decompression alone and decompression plus fusion for LSS have been published. Most of the studies concluded that decompression plus fusion had better clinical outcomes compared with decompression alone. However, in 2016, two randomized control trials (RCT) about LSS were published in the New England Journal of Medicine (NEJM) and raised some serious questions. The results of both studies showed that fusion did not have much additional value for patients with stable LSS, and moreover, it might be regard as an overcautious and unnecessary treatment, which were contradictory to most of the previous studies.

Over the past few years, minimally invasive spine surgery (MISS) has been improving rapidly due to the development of related instruments, more experienced surgeons, and patients' demands. Compared with open spine surgery, MISS has already proved to be associated with less surgical trauma and rapid recovery with similar clinical outcomes. Minimally invasive spinal decompression (MIS-D) and minimally invasive spinal decompression and fusion (MIS-TLIF) have been performed widely for the treatment of LSS. However, there is no previous study comparing MIS-D to MIS-TLIF in terms of clinical outcomes, complications, reoperations, and other perioperative data. Therefore, a randomized controlled trial comparing these 2 common MISS techniques is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Intermittent claudication with pain or numbness or weakness of lower limb(s) with or without low back pain
* An imaging study (MRI or CT) showing single level lumbar spinal stenosis

Exclusion Criteria:

* Insufficient conservative treatment (6 weeks)
* Cauda equina syndrome or progressive neurologic deficit requiring urgent surgical intervention
* Previous spinal surgery
* Other comorbid conditions that contraindicating surgery
* Possible pregnancy that contraindicating radiological examination
* Age less than 18 years old
* Combination with 2°spondylolisthesis or segmental instability (slip distance >4mm or angle change >10° in dynamic plain film)
* Combination with other spinal disorder requiring advanced surgery (such as lumbar stenosis, spondylolisthesis, deformity, fracture, infection, tumor and so on)
* Equal to or more than two responsible level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change in Oswestry Disability Index (ODI) score from baseline | preoperatively and 2 month, 6 months, 1 year，2 years and 5 years postoperatively
  The Oswestry Disability Index (ODI) is widely used to assess chronic low back pain. It contains ten sections including pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and traveling. The ODI is ranging from 0 to 100, with higher scores indicating more disability related to pain.

SECONDARY OUTCOMES:
change in European Quality of Life-5 Dimensions (EQ-5D) from baseline | preoperatively and 2 month, 6 months, 1 year，2 years and 5 years postoperatively
  The EQ-5D is a widely used instrument to assess health-related quality of life. Five questions(Mobility, Self-care, activities of daily living, Pain and Anxiety) are categorical (1-3 scale) and one question is on interval level (0-100).The EQ-5D is ranging from 0 to 1, with a higher score indicating better quality of life.
change in visual analog scales (VAS) from baseline | preoperatively and 2 month, 6 months, 1 year，2 years and 5 years postoperatively
  The VAS score is commonly used for pain assessment, which is ranging from 0 to 10, with higher scores indicating more severe pain
MacNab criteria | 2 month, 6 months, 1 year，2 years and 5 years postoperatively
  The patient is asked to rate his level of well-being, generally after surgery. The patient choose one of the four: Excellent, Good, Fair, Poor.

IPD SHARING:
Plan to Share IPD: No